CLINICAL TRIAL: NCT06500455
Title: Phase III Trial of Single Fraction Stereotactic Radiosurgery (SRS) Versus Fractionated SRS (FSRS) for Intact Brain Metastases
Brief Title: Testing Longer Duration Radiation Therapy Versus the Usual Radiation Therapy in Patients With Cancer That Has Spread to the Brain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN013; NCI-2024-04812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN013 (Other: NRG Oncology); NRG-BN013 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Digestive System Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Renal Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Neoplasm Metastasis; Melanoma; Carcinoma, Renal Cell; Lung Neoplasms | interventions — Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (SRS) (Active Comparator): Patients undergo SRS over 30-90 minutes for 1 fraction on study. Additionally, patients undergo CT and MRI on study.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Radiation: Stereotactic Radiosurgery
- ARM II (FSRS) (Experimental): Patients undergo FSRS over 30-90 minutes for 3 fractions on study. Additionally, patients undergo CT and MRI on study.
  Interventions: Procedure: Computed Tomography; Radiation: Fractionated Stereotactic Radiation Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: Fractionated Stereotactic Radiation Therapy — Undergo FSRS
  Other Names: Fractionated Stereotactic Radiotherapy
  Arms: ARM II (FSRS)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: ARM I (SRS)

SUMMARY:
This phase III trial compares the effectiveness of fractionated stereotactic radiosurgery (FSRS) to usual care stereotactic radiosurgery (SRS) in treating patients with cancer that has spread from where it first started to the brain. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. FSRS delivers a high dose of radiation to the tumor over 3 treatments. SRS is a type of external radiation therapy that uses special equipment to position the patient and precisely give a single large dose of radiation to a tumor. FSRS may be more effective compared to SRS in treating patients with cancer that has spread to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the time to local failure is improved with FSRS compared to SRS in patients with intact (i.e., unresected) brain metastases.

SECONDARY OBJECTIVES:

I. To compare time to intracranial progression-free survival between FSRS and SRS.

II. To compare overall survival between FSRS and SRS. III. To determine if the time to local failure is improved with FSRS compared to SRS, as evaluated by central review of imaging.

IV. To evaluate if there is any difference in central nervous system (CNS) failure patterns (local versus [vs.] distant brain failure vs. both) in patients who receive FSRS compared to patients who receive SRS.

V. To compare the rates of radiation necrosis in patients who receive FSRS vs. SRS.

VI. To compare the time to salvage whole brain radiation therapy (WBRT) between patients who receive FSRS and those who receive SRS.

VII. To compare the rates of post-treatment adverse events associated with FSRS and SRS.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo SRS over 30-90 minutes for 1 fraction on study. Additionally, patients undergo computed tomography (CT) and magnetic resonance imaging (MRI) on study.

ARM II: Patients undergo FSRS over 30-90 minutes for 3 fractions on study. Additionally, patients undergo CT and MRI on study.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of one of the following solid tumor malignancies within 5 years prior to registration:

  * Non-small cell lung cancer
  * Melanoma
  * Breast cancer
  * Renal cell carcinoma
  * Gastrointestinal cancer
  * If the original histologic proof of malignancy is greater than 5 years, then more recent pathologic confirmation (e.g., from a systemic site or brain metastasis) or unequivocal imaging confirmation of extracranial metastatic disease (e.g. CT of the chest/abdomen/pelvis, positron emission tomography [PET]/CT, etc.) is required
* Patients must have at least 1 and up to 8 total intact brain metastases detected on a contrast-enhanced MRI performed ≤ 21 days prior to registration
* At least 1 of the up to 8 lesions must be a study eligible lesion, defined as lesion with a maximum diameter as measured on any orthogonal plane (axial, sagittal, coronal) of ≥ 1.0 cm and ≤ 3.0 cm
* All brain metastases must be located outside of the brainstem and ≥ 5 mm from the optic nerves or optic chiasm and ≤ 3.0 cm in maximum dimension

  * Note: brainstem metastases per the MRI within 21 days of registration are an exclusion criterion; however, if the MRI used for treatment planning performed within 7 days of SRS/FSRS reveals a brainstem metastasis, the patient remains eligible if the patient is considered an appropriate radiosurgery candidate per the local investigator
* Patients must have a diagnosis-specific graded prognostic assessment ≥ 1.5
* No more than 2 lesions planned for resection if clinically indicated
* No known leptomeningeal disease (LMD)

  * Note: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive cerebrospinal fluid (CSF) cytology and/or unequivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In that patient, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion
* Age ≥ 18 years
* Karnofsky performance status (KPS) ≥ 60
* Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* No prior radiotherapy to the brain (partial or whole brain irradiation, SRS, FSRS, or prophylactic cranial irradiation [PCI])
* New York Heart Association Functional Classification II or better (NYHA Functional Classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification)
* No active infection currently requiring intravenous (IV) antibiotic management
* No hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* No chronic obstructive pulmonary disease exacerbation or other acute respiratory illness precluding study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to local failure | From randomization (with the treatment planning magnetic resonance imaging as the 'baseline' for purposes of disease assessment) to local tumor progression of any study lesion(s), assessed up to 5 years
  The time to local failure will be evaluated at a per-patient level. The cause-specific hazard ratio will be estimated in a Cox proportional hazards (PH) model adjusting for patients and disease characteristics. The Cox PH model will be the principle approach. The cumulative incidence function estimator will also be used to estimate the rate of local failure in the presence of competing event of deaths in the two arms separately. A complementary analysis will involve Gray's test to evaluate the difference in the distribution of local failure between treatment arms. These results will be interpreted in light of the competing deaths.

SECONDARY OUTCOMES:
Intracranial progression-free survival (IPFS) | From the date of randomization until intracranial progression (local or distant intracranial) or death from any cause, whichever occurs first, assessed up to 5 years
  IPFS will consist of estimation of its distribution for each treatment arm via the Kaplan-Meier method and a stratified log-rank test. Statistical power will depend on the total IPFS events accumulated at trial end.
Overall survival | From the date of randomization until death from any cause, assessed up to 5 years
  Will consist of estimation of its distribution for each treatment arm via the Kaplan-Meier method and a stratified log-rank test. Reasons for death (e.g. due to neurological cause [any central nervous system event such as an intracranial mass, hemorrhage, or hydrocephalus] or non-neurological cause) will be recorded.
Time to radiation necrosis (TTRN) | From randomization until radiation necrosis, assessed up to 5 years
  The rate of radiation necrosis will be compared in patients who receive fractionated stereotactic radiosurgery to patients who receive stereotactic radiosurgery. The primary comparison of treatment effect on TTRN will be based on testing the cause-specific hazard ratio (CHR) in a univariate Cox proportional hazards model. Additional supplementary analyses will include estimating the cause specific ratio in a Cox proportional hazards model adjusting for patients and disease characteristics (e.g. stratification randomization factors) and estimating the median TTRN via the cumulative incidence function estimator (Korn 1992). The Gray's test will also be used to evaluate the difference in the distribution of TTRN between treatment arms (Gray 1988).
Time to whole brain radiation therapy (WBRT) | Up to 5 years
  Analysis of time to WBRT will consist of estimation of its distribution for each treatment arm via the Kaplan-Meier method and a stratified log-rank test. For patients who die prior to WBRT, time to WBRT will be censored at time of death.
Incidence of adverse events (AEs) | Up to 2 years from start of radiation treatment
  AEs will be graded according to Common Terminology Criteria in Adverse Events version 5.0. Comprehensive summaries of all AEs by treatment arm will be generated and examined. Counts and frequencies of worst AE per patients will be presented overall and by AE type category, separately by assigned treatment group. The proportion of patients with at least one grade 3 or higher AE will be compared between arms. Frequencies for specific potentially treatment related AEs where grade 3 or higher events are noted may be compared. Any frequencies to be tested will be evaluated using the chi-square or exact test as appropriate, with two-sided significance level of 0.05.

OTHER OUTCOMES:
Time to local failure | Up to 5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% confidence interval will be provided by sex, race, and ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Rupesh R Kotecha, Principal Investigator — NRG Oncology
Locations (242):
- United States (239):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Providence Queen of The Valley, Napa, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope South Bay, Torrance, California
  - City of Hope Upland, Upland, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - NRG Oncology, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec, Canada
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Cork Radiation Oncology Associates Limited, Cork, Ireland